CLINICAL TRIAL: NCT00954824
Title: Inflammation and the Metabolic Syndrome in Humans
Acronym: LPS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 706771; 1R01HL073278-01 (NIH)
Record Dates: First submitted 2009-08-05; First posted 2009-08-07 (Estimated); Results first posted 2016-01-28 (Estimated); Last update posted 2017-03-30 (Actual); Status verified 2017-03

CONDITIONS: Metabolic Syndrome X
MeSH Terms: conditions — Metabolic Syndrome | interventions — Endotoxins; Lipopolysaccharides

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Endotoxin (LPS) (Experimental): Single administration low-dose (3 ng/kg) endotoxin (LPS).
  Interventions: Biological: Endotoxin (LPS)

INTERVENTIONS:
Biological: Endotoxin (LPS) — Single administration low-dose (3 ng/kg) endotoxin (LPS).
  Other Names: LPS

SUMMARY:
People who are overweight are at increased risk of heart disease. Being overweight and having heart disease are linked in that both involve inflammation. Inflammation refers to the body's first line of defense against infection and injury. Metabolic changes in cholesterol, triglycerides (fat in the blood) and sugar in the blood caused by inflammation are similar to that in some people who are overweight. The investigators wish to examine the effects of inflammation on these metabolic changes that may lead to heart disease.

DETAILED DESCRIPTION:
This study is a single site, open-label, "baseline-controlled" (pre LPS saline period) study examining the pro-atherosclerotic metabolic responses and safety responses to a single administration low-dose (3 ng/kg) endotoxin (LPS) in 20 additional non-metabolic syndrome participants: 10 healthy overweight and 10 healthy lean counterparts (20 non-metabolic syndrome participants were studies in first phase), and 40 subjects with the metabolic syndrome. We are continuing to use an approach whereby "metabolic syndrome" subjects will be recruited to have key metabolic syndrome abnormalities that are sensitive to insulin resistance compared to the non-metabolic syndrome groups, although all of these "metabolic syndrome" subjects may not fulfill traditional NCEP criteria for the syndrome.

ELIGIBILITY:
Inclusion Criteria:

1. Men and non-pregnant/lactating women between the ages of 18 and 40
2. Subjects must be able to give written informed consent and willing to comply with all study-related procedures.
3. BMI >18 and < 24 and BIA < 15% fat for men, < 25% fat for women, and do not have diagnosis of NCEP metabolic syndrome as defined below, OR
4. BMI > 26 but < 30 and BIA > 15% fat for men, > 25% fat for women, do not have diagnosis of NCEP metabolic syndrome, OR
5. BMI >18 and < 30 and have metabolic syndrome abnormalities as defined below. The modified NCEP Metabolic Syndrome criteria are as follows

   * abdominal obesity, waist circumference: men >= 37 in (94 cm), women >= 31 in (80 cm)
   * fasting triglycerides > 150 mg/dL
   * HDL cholesterol < 40 mg/dL for men; HDL cholesterol < 50 mg/dL for women
   * Blood pressure > 130/ >85 mmHg in untreated patients
   * Fasting glucose > 100 mg/dL, but less than 126 mg/dL
6. For inclusion in "metabolic syndrome" group, the following additional criteria must be fulfilled:

   * Three or more of the NCEP criteria defined above. OR
   * Two or more of the NCEP criteria AND TG/HDL ratio > 3.0.

Exclusion Criteria:

1. Known atherosclerotic cardiovascular disease, including coronary disease, cerebrovascular disease, or peripheral vascular disease.
2. History of diabetes mellitus.
3. A plasma glucose greater than 200 mg/dL at the 2 hour blood draw of the oral glucose tolerance test.
4. History of a non-skin malignancy within the previous 5 years.
5. Renal insufficiency as defined by creatinine >= 1.5 mg/dl at visit 1 (grade 1 of NIH's Common Toxicity Criteria (CTC), version 2.0, 4/30/99).
6. History of liver disease or ALT, AST, ALK Phosphatase or Gamma GT above normal limits as defined by HUP William Pepper Clinical Laboratory at visit 1.
7. Elevated (> 1.5x ULN; grade 1, CTC, 4/30/99) Total Bilirubin or LDH at visit 1.
8. Men who consume > 14 alcoholic drinks per week or > 4 alcoholic drinks per occasion (AMA/NIAAA criteria for "at risk" usage levels).
9. Women who consume > 7 alcoholic drinks per week or > 3 alcoholic drinks per occasion (AMA/NIAAA criteria for "at risk" usage levels).
10. Total white blood cell count below normal limits as defined at HUP William Pepper Clinical Laboratory prior to the baseline visit.
11. Hemoglobin below normal limits (gender specific) as defined at HUP William Pepper Clinical Laboratory prior to the baseline visit.
12. Any medical condition or abnormal laboratory value that is judged clinically significant by an investigator.
13. Any major active rheumatologic, pulmonary, or dermatologic disease or inflammatory condition or minor active infection.
14. History of HIV positive.
15. First degree family history of premature cardiovascular disease event (father or brother if diagnosed at before 55 years of age; mother or sister if diagnosed before 65 years of age).
16. Patients who have undergone any organ transplant.
17. Individuals who currently use tobacco products or have done so in the previous 30 days.
18. Treatment with aspirin, NSAIDs, COX-2 inhibitors, steroids or other immunomodulatory therapy 2 weeks prior to the screening visit
19. Treatment with statins, fibrates or niacin 4 weeks prior to the screening visit.
20. Current daily use of Vitamin C > 1000 mg, Beta carotene > 1000 IU, vitamin A > 5000 IU, vitamin E > 400 IU, and selenium > 200 mcg.
21. Positive urine pregnancy at the screening visit.
22. Participation in another clinical trial within the previous 6 weeks prior to the screening visit.
23. Poorly controlled blood pressure (BP > 160/100) or on any anti-hypertensive medications.
24. For subjects in non-metabolic syndrome groups; a diagnosis of metabolic syndrome using NCEP ATPIII criteria.
25. For subjects in "metabolic syndrome" group; an abnormal Bruce protocol cardiac exercise stress test.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2003-08; Primary Completion 2007-11 (Actual); Study Completion 2007-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Muredach P. Reilly, MB, MSCE, Principal Investigator — University of Pennsylvania
Locations (1):
- Clinical and Translational Research Center, Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Background] Anderson PD, Mehta NN, Wolfe ML, Hinkle CC, Pruscino L, Comiskey LL, Tabita-Martinez J, Sellers KF, Rickels MR, Ahima RS, Reilly MP. Innate immunity modulates adipokines in humans. J Clin Endocrinol Metab. 2007 Jun;92(6):2272-9. doi: 10.1210/jc.2006-2545. Epub 2007 Mar 20. PMID 17374708
- [Background] Heffron SP, Parastatidis I, Cuchel M, Wolfe ML, Tadesse MG, Mohler ER 3rd, Ischiropoulos H, Rader DJ, Reilly MP. Inflammation induces fibrinogen nitration in experimental human endotoxemia. Free Radic Biol Med. 2009 Oct 15;47(8):1140-6. doi: 10.1016/j.freeradbiomed.2009.07.025. Epub 2009 Jul 22. PMID 19631267
- [Background] Shah R, Lu Y, Hinkle CC, McGillicuddy FC, Kim R, Hannenhalli S, Cappola TP, Heffron S, Wang X, Mehta NN, Putt M, Reilly MP. Gene profiling of human adipose tissue during evoked inflammation in vivo. Diabetes. 2009 Oct;58(10):2211-9. doi: 10.2337/db09-0256. Epub 2009 Jul 6. PMID 19581417
- [Background] McGillicuddy FC, de la Llera Moya M, Hinkle CC, Joshi MR, Chiquoine EH, Billheimer JT, Rothblat GH, Reilly MP. Inflammation impairs reverse cholesterol transport in vivo. Circulation. 2009 Mar 3;119(8):1135-45. doi: 10.1161/CIRCULATIONAHA.108.810721. Epub 2009 Feb 16. PMID 19221221
- [Background] Badellino KO, Wolfe ML, Reilly MP, Rader DJ. Endothelial lipase is increased in vivo by inflammation in humans. Circulation. 2008 Feb 5;117(5):678-85. doi: 10.1161/CIRCULATIONAHA.107.707349. Epub 2008 Jan 22. PMID 18212282
- [Background] Song WL, Wang M, Ricciotti E, Fries S, Yu Y, Grosser T, Reilly M, Lawson JA, FitzGerald GA. Tetranor PGDM, an abundant urinary metabolite reflects biosynthesis of prostaglandin D2 in mice and humans. J Biol Chem. 2008 Jan 11;283(2):1179-88. doi: 10.1074/jbc.M706839200. Epub 2007 Nov 8. PMID 17993463
- [Background] Lehrke M, Millington SC, Lefterova M, Cumaranatunge RG, Szapary P, Wilensky R, Rader DJ, Lazar MA, Reilly MP. CXCL16 is a marker of inflammation, atherosclerosis, and acute coronary syndromes in humans. J Am Coll Cardiol. 2007 Jan 30;49(4):442-9. doi: 10.1016/j.jacc.2006.09.034. Epub 2007 Jan 12. PMID 17258089
- [Background] Reilly MP, Lehrke M, Wolfe ML, Rohatgi A, Lazar MA, Rader DJ. Resistin is an inflammatory marker of atherosclerosis in humans. Circulation. 2005 Feb 22;111(7):932-9. doi: 10.1161/01.CIR.0000155620.10387.43. Epub 2005 Feb 14. PMID 15710760
- [Background] Lehrke M, Reilly MP, Millington SC, Iqbal N, Rader DJ, Lazar MA. An inflammatory cascade leading to hyperresistinemia in humans. PLoS Med. 2004 Nov;1(2):e45. doi: 10.1371/journal.pmed.0010045. Epub 2004 Nov 30. PMID 15578112

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Non-tobacco using individuals between ages 18-40 in 2 groups- with metabolic syndrome (having 3 of 5 criteria) and non-metabolic syndrome.
Period: Overall Study
Arm/Group | Endotoxin (LPS)
Started | 100
Completed | 50
Not Completed | 50

BASELINE CHARACTERISTICS:
Arm/Group | Endotoxin (LPS)
Number analyzed (Participants) | 50
Age, Continuous [Mean (Full Range); unit: years] | 25.6 [19 to 40]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23
  Male | 27

OUTCOME MEASURES:

1. Primary Outcome: The Primary Outcome Measure is Plasma Levels of TNF Alpha.
Time Frame: 24 hours
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Endotoxin (LPS)
Number analyzed (Participants) | 20
ng/mL | 507 (251)

ADVERSE EVENTS:
Arm/Group | Endotoxin (LPS)
Serious Adverse Events (participants affected / at risk) | 0/100
Other Adverse Events (participants affected / at risk) | 32/100
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Endotoxin (LPS) (N=100)
Vomitting (Gastrointestinal disorders) | 16 (24)
rigors (Musculoskeletal and connective tissue disorders) | 4 (4)
HR < 50bpm (Cardiac disorders) | 4 (4)
Vagal reaction (Nervous system disorders) | 4 (4) — also termed vaso-vagal events or syncope
superficial thrombophlebitis (Vascular disorders) | 4 (4) — from IV site used over the course of inpatient visit

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes